CLINICAL TRIAL: NCT07125144
Title: Piloting a Culturally Adapted Multilevel Suicide Prevention Intervention in Schools for Black Youth and Their Families
Brief Title: Piloting a Culturally Adapted Suicide Prevention for Black Students in Chicago
Acronym: SP-BSC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Janelle Goodwill, Neubauer Family Assistant Professor, University of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH129789 (NIH); R34MH129789 (NIH)
Record Dates: First submitted 2025-08-04; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Suicide; Suicidal Ideation; Suicide Attempt
Keywords: Black; youth; suicide; suicide prevention; intervention; Signs of Suicide; Cultural Adaptation; Chicago; African American; Adolescent
MeSH Terms: conditions — Suicide; Suicidal Ideation; Suicide, Attempted; Suicide Prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard/Existing Intervention (Active Comparator): Students attending schools assigned to the Standard/Existing Intervention condition will receive the existing Signs of Suicide intervention.
  Interventions: Behavioral: Signs of Suicide: Standard/Existing
- Culturally Adapted Intervention (Experimental): Students attending schools assigned to the Culturally Adapted Intervention condition will receive a new culturally adapted intervention developed for this study.
  Interventions: Behavioral: Black Youth Suicide Prevention in Chicago

INTERVENTIONS:
Behavioral: Black Youth Suicide Prevention in Chicago — The Culturally Adapted intervention uses intervention video content that specifically addresses topics that shape Black youth's psychological wellbeing and development. The goal of this intervention is to share suicide prevention information in ways that are culturally responsive and attentive to the specific needs of Black adolescents.
  Arms: Culturally Adapted Intervention
Behavioral: Signs of Suicide: Standard/Existing — Students attending schools assigned to the Standard/Existing Intervention condition will receive the Signs of Suicide curriculum.
  Arms: Standard/Existing Intervention

SUMMARY:
Suicide has been the third leading cause of death for Black youth in the U.S since the 1980s and persists as a leading cause of death for Black youth today. For example, in 2018 suicide was reported as the 2nd leading cause of death among Black Americans ages 10 to14 years old. Findings yielded from recent queries indicate that the gap in suicides among Black males and female youth has narrowed in recent years. Despite these disturbing trends, a dearth persists in our understanding of the factors that contribute to and prevent against suicide in Black youth, thus diminishing researchers' ability to effectively detect suicide risk in this particular population. This project aims to redress this gap by proposing the cultural adaptation of an existing suicide prevention intervention, the Signs of Suicide (SOS) prevention program, for Black middle school students. Our team will conduct a pilot randomized controlled trial among a sample of Black middle school students to assess feasibility and

examine underlying mechanisms that contribute to suicidality among Black youth. Intervention content will be adapted to assess how topics of racial identity, racial socialization, and racial discrimination uniquely impact Black youth's mental health experiences and risk for suicide. Measures of suicidal ideation, planning, and attempt will be assessed at pre-test, post-test, and 3-months after the intervention. Findings derived from this project will contribute to public health priorities by offering unique insight into the factors that either prevent or promote suicide among Black youth and could be replicated in other schools serving Black students across the nation.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in 6th, 7th, or 8th grade at a participating school

Exclusion Criteria:

* Not enrolled in 6th, 7th, or 8th grade at a participating school

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation | Baseline, 2 weeks after baseline, 3-months after baseline
  Item that asks students to report if they have seriously considered suicide

SECONDARY OUTCOMES:
Suicide Attempt | Baseline, 2 weeks after baseline, 3-months after baseline
  Item that asks students to report if they have attempted suicide.
Knowledge of Depression and Suicide | Baseline, 2 weeks after baseline, 3-months after baseline
  This scale includes items that assess students' knowledge of depression and suicide risk and warning signs. This is the title of the scale, as used and reported in earlier suicide prevention interventions (Aseltine & DeMartino, 2004; Schilling et al., 2016). Responses are collected using a list of true/false options. The total number of "true" statements represents more accurate knowledge of depression and suicide risk warning signs.
Attitudes Towards Depression and Suicide | Baseline, 2 weeks after baseline, 3-months after baseline
  This scale includes Items that assess students' attitudes towards depression and suicide. This is the title of the scale, as used and reported in earlier suicide prevention interventions (Aseltine & DeMartino, 2004; Schilling et al., 2016). The measure includes a 5-point Likert scale with responses ranging from 1 = "Strongly Disagree" to 5 = "Strongly Agree." Higher scores on this scale represent more adaptive attitudes towards depression and suicide risk.

CONTACTS AND LOCATIONS:
Overall Officials: Janelle R. Goodwill, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Specific data describing participants grade level and scores on primary outcome measures will be made available, per NIMH Data Archive guidelines.
Supporting Information: ICF
Time Frame: Specific data will be submitted to and hosted on the NIMH Data Archive website.
Access Criteria: Specified data will be shared in compliance with NIMH Data Archive guidelines.